CLINICAL TRIAL: NCT04088916
Title: Proviral DNA as a Target for HIV-1 Resistance Analysis
Acronym: HIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, PABLO ANDRES FERRER CAMPOS, Assistant Professor, University of Chile
Other Study IDs: Nº OAIC 986/18
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: HIV/AIDS; HIV Infections; HIV Seropositivity; Viral Infection
Keywords: ADNproviral; HIV; Resistance; genotyping
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; HIV Seropositivity; Virus Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — HIV ADN proviral
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In summary, in this project the investigators propose to study the proviral DNA genotyping to implement a lower cost and wider than the commercial systems currently in use, in order to analyze all HIV genes that are therapeutic targets of antiretroviral drugs. Using HIV proviral DNA we can obtain information for: HIV-1 Viral Tropism, Mutations associated to Integrase Inhibitors, Mutations associated to Transcriptase reverse Inhibitors, Mutations associated to Protease Inhibitors, and Mutations associated to GP41 Inhibitors.

Along with this the investigators propose to validate the proviral DNA as starting material for genotyping which is independent of the patient's viral load and achieve a greater number of patients living with HIV have access to this important test that is essential in monitoring the HIV infection.

3.2 RESEARCH QUESTIONs Is proviral DNA a genetic compartment suitable for carrying out a genotypic resistance test in patients with low or undetectable viral load? Does proviral DNA have the same clinical validity that RNA? 3.3.- HYPOTHESIS A resistance genotyping test carried out by Proviral DNA detects the same mutations associated to resistance that viral RNA.

3.4.- OBJECTIVES: General/Specific General objective Develop a methodology to assess the proviral HIV-1 DNA or RNA as the genetic material for genotyping assays in genes that are targets of pharmacological interest as TR reverse transcriptase and protease (PRO), Integrase or GP41 Inhibitors and HIV tropism. Specific Objectives

1. Carry out genotyping by proviral DNA and compare it with the same genes genotyping performed with viral RNA. 2. Once the correlation between proviral DNA and RNA has shown, standardize a method to use the technique for clinical use in monitoring HIV patients according to each patient's needs. RNA for patients with viral load above 1,000 copies/mL. Proviral DNA for patients with low or undetectable viral load.

DETAILED DESCRIPTION:
A prospective longitudinal observational study, the objective is to observe and describe the prevalence of INRT, INNRT, Protease and INIS mutations detected by proviral DNA in patients with virologic failure and low level viremia.

Inclusion/Exclusion: Our Study will include only patients with HIV that had been confirmed by "Instituto de Salud Pública de Chile" (ISP-Chile). Children less than 18 years are excluded.

Number of Patients: A total of 1,200 patients will be included in a period of three years (Including statistical justification, if appropriate).

1. - Only patients who have signed informed consent will be admitted to our study.
2. - The admitted patients will have a blood sample taken for an HIV genotypic resistance test.
3. - from the clinical record of each patient admitted, some relevant clinical data will be taken to interpret the results such as CD4 T lymphocyte count, Viral Load, date of HIV diagnosis, date of initiation of therapy in addition to number and type of treatments antiretrovirals
4. - By way of genotype control, a second blood sample will be taken every year.

Detailed Description

Detection of Resistance Mutations in Proviral DNA in HIV-1 Infection

Background The genetic test HIV proviral DNA (HPD) for resistance to antiretroviral drugs is very useful to detect mutations in patients under antiretroviral therapy who has failed to achieve undetectable viral loads levels or with low level viremia (LLV).

HPD allows the detection of circulating resistant variants and archived which could not be detected in the plasma.

HPD is independent of the viral load of patients. This makes it very useful for studies of primary resistance as it can detect resistance mutations in recently diagnosed patients with low baseline viral loads (<1,000 copies/mL).

HPD is recommended by the European AIDS Clinical Society EACS for cases where there is not HIV RNA for analysis (Barcelona, October 2015).

HPD is able to analyze resistance to all antiretroviral drugs currently available in the market. Therefore, with the HPD innovation we can carry out the following genetic resistance tests: HIV Tropism (Maraviroc), resistance to Integrase Inhibitors (Dolutegravir) and resistance to Transcriptase reversa/Proteasa (Abacavir).

Size Sample and Methodology

During a period of two years, we will study a population of 1,200 patients. These include all patients we have analyzed in our HIV center until December 2012. The methodology includes nucleic acid extraction, amplification of HIV-1 genes that are targets of therapeutic interest and sequencing by traditional and new generation sequencing methods.

Patient Recruitment: a Total of 1.200 (400 by year)

Obtaining blood samples: two samples: sample to the start and one sample to the end after one year

DNA and viral RNA extraction:

RT-PCR amplification:

Electrophoresis visualization in agarose gels

Sending samples to Macrogen for sequencing services

Automatic sequencing by Sanger method in Macrogen USA

Sequencing by deep sequencing (NGS) in Chile or Macrogen USA

Sequence Analysis

Quality Analysis and assemble of raw sequences in software ReCall

Registry of mutations of clinical interest

Report on resistance to antiretroviral drugs

Biostatistical analysis

Results Report and Publications

Preliminary results Preliminary analysis of 100 patients with viral load <1,000 copies/mL, detected 10% of patients with mutations of resistance to drugs that inhibit reverse transcriptase and viral protease. This valuable information enabled earlier therapeutic intervention by changing the drug scheme before they reach higher levels of viral load with consequent improvement in the clinical management.

Projections Project Due to the success and immediate application of this preliminary study, we believe it become very important to validate this technique as a daily routine genetic testing for HIV clinic patients in the public health system. Permanent financing for this genetic HIV test for HIV proviral DNA should be given by the Ministry of Health, Government of Chile.

In conclusion, at present HPD is very useful tool to study virologic failure and LLV in order to an early change of the antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of HIV

viral load <1.000 copies/mL

under antiretroviral tratment

Exclusion Criteria:

HIV negative

viral load >1.000 copies/mL

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion/Exclusion: Our Study will include only patients with HIV that had been confirmed by "Instituto de Salud Pública de Chile" (ISP-Chile). Children less than 18 years are excluded.
  Number of Patients: A total of 1,200 patients will be included in a period of three years (Including statistical justification, if appropriate)
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-09-08 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Proviral DNA as a Target for HIV-1 Resistance Analysis | 3 years
  Develop a methodology to assess the proviral HIV-1 DNA or RNA as the genetic material for genotyping assays in genes that are targets of pharmacological interest as TR reverse transcriptase and protease (PRO), Integrase or GP41 Inhibitors and HIV tropism

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Ferrer, Dr, Principal Investigator — University of Chile
Locations (2):
- Chile (2):
  - Immunology, HIV and Allergy Section, Santiago, Santiago Metropolitan
  - Molecular Medicine Laboratory, Santiago, Santiago Metropolitan